CLINICAL TRIAL: NCT05662397
Title: An Open Label, Phase 1/2 Study of HST-1011 Given as Monotherapy and in Combination With an Anti-PD1 Antibody in Patients With Advanced Solid Tumors
Brief Title: A Study of HST-1011 Given as Monotherapy and in Combination With an Anti-PD1 Antibody
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: HotSpot Therapeutics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Clin-001
Record Dates: First submitted 2022-12-02; First posted 2022-12-22 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-02

CONDITIONS: Solid Tumor, Adult; Relapsed Cancer; Refractory Cancer
Keywords: CBL-B; anti-PD-(L)1
MeSH Terms: conditions — Recurrence; Neoplasms | interventions — cemiplimab; spartalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- HST-1011 Monotherapy Dose Escalation (Part A1) (Experimental): Multiple dose levels of HST-1011 to be evaluated.
  Interventions: Drug: HST-1011
- HST-1011 Monotherapy Dose Optimization (Part A2) (Experimental): Evaluation of HST-1011 monotherapy dose/dose regimen.
  Interventions: Drug: HST-1011
- HST-1011 Dose Escalation in Combination with cemiplimab (Part B1) (Experimental): Multiple dose levels of HST-1011 to be evaluated in combination with cemiplimab.
  Interventions: Drug: HST-1011; Biological: Cemiplimab
- HST-1011 Dose Optimization in Combination with Cemiplimab (Part B2) (Experimental): Evaluation of HST-1011 in combination with cemiplimab.
  Interventions: Drug: HST-1011; Biological: Cemiplimab

INTERVENTIONS:
Drug: HST-1011 — HST-1011 given orally
  Other Names: CBL-B inhibitor
Biological: Cemiplimab — Cemiplimab administered via intravenous infusion in combination with HST-1011 given orally
  Other Names: anti-PD1 antibody
  Arms: HST-1011 Dose Escalation in Combination with cemiplimab (Part B1); HST-1011 Dose Optimization in Combination with Cemiplimab (Part B2)

SUMMARY:
This is a Phase 1/2 study of HST-1011, a CBL-B inhibitor, being developed for the treatment of patients with advanced solid tumors, who relapsed while on or are refractory to approved anti-PD(L)1 therapies or other standard of care.

DETAILED DESCRIPTION:
This is a Phase 1/2 study of HST-1011, a CBL-B inhibitor, being developed for the treatment of patients with advanced solid tumors, who relapsed while on or are refractory to approved anti-PD(L)1 therapies or other standard of care.

In Phase 1 patients will receive HST-1011 as either monotherapy (Parts A1 and A2) or in combination with the anti-PD1 antibody, cemiplimab (Part B1 and B2).

Part A1 is a monotherapy dose escalation in which cohorts of patients will receive increasing doses of HST-1011. Upon completion of Part A1 dose escalation, an HST-1011 monotherapy dose optimization will commence (Part A2).

Part B1 is a dose escalation of HST-1011 given in combination with the standard dose/regimen of cemiplimab. Dosing in Part B1 may commence prior to the completion of Part A1. Upon completion of Part B1 dose escalation, an HST-1011 dose optimization in combination with cemiplimab will commence (Part B2).

Phase 2 will evaluate the preliminary antitumor activity of HST-1011 in combination with anti-PD(L)1 antibody or other standard of care therapies.

ELIGIBILITY:
Key Inclusion Criteria:

* Patient is at least 18 years of age.
* Patient is capable of understanding and complying with protocol requirements.
* Patient has signed and dated ICF.
* Patient has a histologically confirmed, advanced solid tumor (metastatic, recurrent, and/or unresectable) in one of the following categories: 1) anti-PD-(L)1 relapsed/refractory; 2) platinum-resistant ovarian cancer; 4) anal cancer; 5) rectal cancer; or 6) castration-resistant prostate cancer
* Patient has failed prior standard of care therapies appropriate for their metastatic disease.
* Patient has at least 1 measurable non-central nervous system (CNS) lesions per RECIST 1.1.
* Patient has provided consent for pre- and on-treatment biopsies.
* Eastern Cooperative Performance Status of 0 or 1.

Key Exclusion Criteria:

* Patient has active autoimmune disease or other medical conditions requiring chronic systemic steroid therapy at the time of screening.
* Patient has an unacceptable intolerance to anti-PD-(L)1 monoclonal antibody (Part B Only).
* Patient has previously participated in a clinical study evaluating a CBL-B inhibitor.
* Patients has untreated and/or symptomatic metastatic CNS disease.
* Patient is currently taking any concomitant medications at Screening that have the potential to cause a clinically relevant drug-drug interaction with HST-1011.
* Patients with a history of gastrointestinal disease that may affect absorption of the study drug, or patients who are not able to take oral medications.
* Patient has an active infection requiring systemic therapy.
* Patient has known or suspected infection with SARS-CoV-2 virus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluate the safety and tolerability of escalating doses of single-agent HST-1011 in Part A1 or in combination with cemiplimab in Part B1. | 12 months
  Number of participants with DLTs, with Adverse Events (TEAEs, SAEs), with abnormal clinically significant vital signs, Electrocardiograms (ECGs), with abnormal physical examination findings, and abnormal laboratory test results.
To determine the Recommended Phase 2 Dose (RP2D) and schedule of HST-1011 monotherapy in Part A2 and in combination with cemiplimab in Part B2. | 12 months
  Integration of safety, PD, PK, and preliminary efficacy endpoints.

SECONDARY OUTCOMES:
Evaluate the safety and tolerability of single-agent HST-1011 in Part A2. | 12 months
  Number of participants with Adverse Events (TEAEs, SAEs), with abnormal clinically significant vital signs, Electrocardiograms (ECGs), with abnormal physical examination findings and abnormal laboratory test results.
Measurement of plasma concentrations of HST-1011 after monotherapy in Part A1 and Part A2 or in combination with cemiplimab in Part B to derive summary pharmacokinetic (PK) parameters including Tmax, Cmax, AUC0-last, Ctrough. | 12 months
  Characterize pharmacokinetic parameters including Tmax, Cmax, AUC0-last, Ctrough after oral administration of HST-1011 or combination of orally administered HST-1011 and IV infused cemiplimab.
Characterize the concentration of peripheral blood cytokines/chemokines following HST-1011 monotherapy Part A1 and Part A2, or in combination with cemiplimab in Part B1. | 12 months
  Measure of peripheral pharmacodynamic (PD) markers after oral administration of HST-1011 or combination of orally administered HST-1011 and IV infused cemiplimab.
Characterize global gene expression profiles following HST-1011 monotherapy Part A1 and Part A2, or in combination with cemiplimab in Part B1 and Part B2. | 12 months
  Measure of peripheral pharmacodynamic (PD) markers after oral administration of HST-1011 or combination of orally administered HST-1011 and IV infused cemiplimab.
Evaluate intratumoral gene expression changes of single-agent HST-1011 in Part A2 and in combination with cemiplimab in Part B2. | 12 months
  Measure of intratumoral pharmacodynamic (PD) markers after oral administration of HST-1011 alone and in combination with cemplimab.
Overall Response Rate (ORR) following HST-1011 monotherapy Part A1 and Part A2, or in combination with cemiplimab in Part B1 and Part B2. | 12 months
  Defined as the percentage of subjects who have a complete response (CR) or partial response (PR), as determined according to RECIST v1.1, or to PCWG for CRPC, if applicable.
Duration of response (DOR) of single-agent HST-1011 in Part A2, or in combination with cemiplimab in Part B2. | 12 months
  Defined as the time from when the criteria for RECIST 1.1, or to PCWG for CRPC, if applicable, CR or PR (whichever is recorded first) was first met until the date when progressive disease is documented.
Disease Control Rate (DCR) of single-agent HST-1011 in Part A2, or in combination with cemiplimab in Part B2. | 12 months
  Defined as the percentage of subjects who have a CR or PR or stable disease (SD), as determined according to RECIST v1.1, or to PCWG for CRPC, if applicable.
Progression Free Survival (PFS) of single-agent HST-1011 in Part A2, or in combination with cemiplimab in Part B2. | 12 months
  Defined as the time from first treatment to first occurrence of progressive disease or death from any cause.
Overall Survival (OS) of single-agent HST-1011 in Part A2, or in combination with cemiplimab in Part B. | 12 months
  Defined as the time from first treatment to death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Alison O'Neill, MD, Study Director — HotSpot Therapeutics, Inc
Locations (14):
- United States (8):
  - Florida Cancer Specialists, Sarasota, Florida
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Montefiore Einstein Comprehensive Cancer Center, The Bronx, New York
  - Providence Cancer Institute of Oregon, Portland, Oregon
  - Abramson Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh (UPMC), Hillman Cancer Center, Pittsburgh, Pennsylvania
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
- Canada (2):
  - University of Ottawa, Ottawa, Ontario
  - Princess Margaret Cancer Center, Toronto, Ontario
- Spain (4):
  - NEXT Oncology Barcelona IOB Hospital Quirónsalud, Barcelona
  - Clínica Universidad de Navarra, Madrid
  - NEXT Oncology Hospital Universitario Quirónsalud Madrid, Madrid
  - Clínica Universidad de Navarra (Pamplona), Pamplona

IPD SHARING:
Plan to Share IPD: No